CLINICAL TRIAL: NCT02648191
Title: Preoperative Treatment With Noninvasive Intra-auricular Vagus Nerve Stimulation Pending Bariatric Surgery. A Randomized, Controlled, Double-blind Trial
Brief Title: Preoperative Treatment With Noninvasive Intra-auricular Vagus Nerve Stimulation Pending Bariatric Surgery
Acronym: OBESITE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion and departure of the investigator
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1508013; 2015-A00253-46 (Other: ANSM)
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Obesity; Bariatric Surgery; No invasive intra-auricular vagus nerve stimulation; Weight loss; Autonomic nervous system
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active stimulation (Experimental)
  Interventions: Device: NeuroCoach II Stim
- Inactive stimulation (Sham Comparator)
  Interventions: Device: NeuroCoach II Stim

INTERVENTIONS:
Device: NeuroCoach II Stim — A noninvasive vagus nerve stimulator consists of two components. An electrode is placed in the left ear concha and will be used by the patient for 4-5 hours per day in segments of 1 hour minimum.
  For this intervention, the stimulations are active.
  Other Names: NeuroCoach II Stim, NBA Techno, France
  Arms: Active stimulation
Device: NeuroCoach II Stim — A noninvasive vagus nerve stimulator consists of two components. An electrode is placed in the left ear concha and will be used by the patient for 4-5 hours per day in segments of 1 hour minimum.
  For this intervention, the stimulations are inactive.
  Other Names: NeuroCoach II Stim, NBA Techno, France
  Arms: Inactive stimulation

SUMMARY:
Faced with the current obesity epidemic, new avenues of research into effective weight loss must be developed.

Among the possible actions on obesity, vagus nerve stimulation has been shown in several studies to be effective in treating epilepsy or depression, at the same time inducing weight loss in those patients. Vagus nerve stimulation has also shown to be effective on weight loss in experimental animal studies. Vagus nerve stimulation has never been attempted in obese patients awaiting bariatric surgery.

DETAILED DESCRIPTION:
The primary objective is to demonstrate the benefit of transcutaneous vagus nerve stimulation in obese subjects awaiting surgery. Secondary objectives include, among others, the risk factors related to obesity, systemic micro-inflammation, insulin and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Any obese patient consulting for bariatric surgery with BMI ≥ 35 and comorbidities or with BMI ≥ 40
* Consent Form signed

Exclusion Criteria:

* Permanent atrial fibrillation
* Patient on treatment that could influence measurement of Autonomic Nervus System (ANS) activity (eg. anti-arrhythmics).
* For patients previously operated (by any technique), an interval of at least 6 months since the surgery must be observed
* Pacemaker
* Serious cardiac pathology
* History of myocardial infarction
* History of Stroke
* Severe respiratory insufficiency
* Allergy in the Rhodium and in the gold
* Surgery of the vagus nerve
* Pregnant patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Weight | at 6 months
  the weight (kg) is measured after 6 months of noninvasive stimulation.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | at 3, 6, 9 and 12 months
  HRV is measured by a 24H-Holter Electrocardiography (ECG). It is a composite outcome :
  * the standard deviation of NN intervals (SDNN)
  * the proportion of number of pairs of successive NNs that differ by more than 50 ms, divided by total number of NNs (pNN50)
  * high frequency (HF)
  * low frequency (LF)
  * very low frequency (VLF)
Systemic inflammation | at 3, 6, 9 and 12 months
  Markers of systemic inflammation will be measured on centrifuged serum for C-reactive protein (CRP) and by immuno microassay using the Luminex method for InterLeukin (IL)-6 and IL-17.
Apnea-hypopnea index (AHI) | at 3, 6, 9 and 12 months
  AHI is analyzed by a polysomnography in an outpatient setting.
Patient Health Questionnaire-9 (PHQ-9) | at 3, 6, 9 and 12 months
  It is a anxiety scale
Blood pressure | at 1, 3, 6, 9 and 12 months
Octanoylated ghrelin hormone | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Glucagon-like peptide-1 hormone (GLP1) | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Peptide tyrosine tyrosine hormone (PYY) | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Lipide profile (Cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglyceride) | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Serum insulin level | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Glycemia | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Glycated hemoglobin | at 3, 6, 9 and 12 months
  Patients will be subjected to blood samplings
Adverse effects | at 12 months
  Local and systemic adverse effects will be described at each consultation. In particular, patients will be informed that they can call the investigator if they have any questions or to report any effects that seem unusual.

CONTACTS AND LOCATIONS:
Overall Officials: Radwan KASSIR, MD, Principal Investigator — CHU de St Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No